CLINICAL TRIAL: NCT06908876
Title: A Randomized, Double-maskedblind, Activity-controlled Phase II Clinical Study to Evaluateing the Efficacy and Safety of Intravitreal Injection of IBI302 in Patients With Diabetic Macular Edema（DME） Subjects
Brief Title: A Study to Evaluate the Efficacy and Safety of IBI302 inSubjects With Diabetic Macular Edema（DME）
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics Technology Limited (Shanghai R&D Center) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIBI302B202
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Macular Oedema
MeSH Terms: interventions — IBI302; faricimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IBI302 Dose 8mg (Experimental): Drug: IBI302 8mg/eye; Intraocularinjection
  Interventions: Biological: IBI302
- Faricimab (Active Comparator): Drug: Faricimab 6mg/eye; Intraocularinjection
  Interventions: Drug: Faricimab
- IBI302 Dose 4mg (Experimental): Drug: IBI302 4mg/eye; Intraocularinjection
  Interventions: Biological: IBI302

INTERVENTIONS:
Biological: IBI302 — 4 mg IBI302 will be administered by intravitreal injection into the study eye once every 4 weeks for 3 consecutive months, followed by Pro re nata (PRN) regimen.
  Arms: IBI302 Dose 4mg
Biological: IBI302 — 8 mg IBI302 will be administered by intravitreal injection into the study eye once every 4 weeks for 3 consecutive months, followed by PRN regimen.
  Arms: IBI302 Dose 8mg
Drug: Faricimab — 6 mg faricimab will be administered by intravitreal injection into the study eye once every 4 weeks for 4 consecutive months, followed by PRN regimen.
  Arms: Faricimab

SUMMARY:
The study is designed for multi-center,randomized,double-masked,active-contralledstudy to evaluate effective and security of intravitrealinjection of IBI302 in subjects with Diabetic Macular Oedema.

ELIGIBILITY:
Inclusion criteria：

* Informed Consent Form (ICF) must be signed before participating in the study, compliance is good, and willing to complete the visit as planned;
* Subjects aged 18-80 years (inclusive) at the time of screening, and diagnosed with type I or type II diabetes;
* DME involved the macular fovea at screening;
* CST≥320 μm as confirmed by OCT in the study eye at screening.
* At baseline, visual acuity loss in the study eye due to DME with BCVA ranging from 19 to 78 ETDRS letters (inclusive);
* Currently use of insulin, or other injectable drugs, or oral hypoglycemic agents to treat diabetes, HbA1c ≤10% at screening;

Exclusion criteria： Eye disease

* High-risk PDR in the study eye;
* Dense hard exudation that destroyed the fovea structure of the macula in the study eye;
* Iris neovascularization in the study eye;
* Other systemic/ocular disease associated with the study eye may cause subjects fail to respond to study treatment or confuse the interpretation of study findings;
* Uncontrolled glaucoma in the study eye; Eye treatment
* Any previous treatment with IBI302 in the study eye before baseline;
* Intravitreal injection of anti-VEGF or anti-complement agents in the study eye within 90 days prior to baseline;
* Panretinal photocoagulation or macular laser (focal, grid or micropulse) in the study eye within 90 days prior to baseline;
* Cataract surgery was performed in the study eye within 90 days prior to baseline;
* YAG laser capsulotomy or YAG laser peripheral iridotomy were performed in the study eye within 90 days prior to baseline.
* Any other intraocular surgery (eg, corneal transplantation, glaucoma filtration, pars plana vitrectomy, or radiotherapy) Systemic diseases/treatments
* Currently untreated diabetes mellitus or previously untreated patients who initiated oral or injectable antidiabetic medication <90 days prior to administration.
* Uncontrolled hypertension.
* Systemic use of anti-VEGF or anti-complement agents within 90 days prior to baseline
* The presence of any other pre-existing disease, metabolic disorder, abnormal results on a physical examination or clinical laboratory examination that may reasonably be suspected of causing contraindications with the investigational drug, or affecting the interpretation of study results, or placing subjects at high risk of treatment complications (e.g., coagulation dysfunction, history of acute cardiovascular and cerebrovascular disease, history of treated or untreated malignancies within the past 5 years, etc.);
* Systemic treatment for suspected or active systemic infection (e.g., tuberculosis, hepatitis B, hepatitis C, etc.);
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
BCVA change from baseline | From Baseline through At Week 16
  Change from baseline in BCVA as measured on The BCVA is measured by Early Treatment Diabetic Retinopathy Study (ETDRS) chart at week 16.

SECONDARY OUTCOMES:
The proportion of patients with an ≥ 2-step DRSS improvement | At Week 16 and 36
  DRSS level is evaluated by color fundus photography (CFP).
The proportion of patients with PDR | The proportion of patients with PDR
  The presence of PDR is evaluated by CFP.
The proportion of new developed PDR | At Week 16 and 36
  The presence of new developed PDR is evaluated by CFP.
Change from baseline in BCVA over time | From Baseline through Week 36
  Change from baseline in BCVA as measured on ETDRS chart
The proportion of patients with CST < 320 μm over time | From Baseline through Week 36
  CST is measured by Optical coherence tomography (OCT).
AEs over time | From Baseline through Week 36
  All AEs were recorded and the investigator made an assessment on severity and causality of each AE.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General hospital, Shanghai, Shanghai Municipality, China